CLINICAL TRIAL: NCT06747416
Title: A Phase II Multicenter, Open Label Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, Pharmacodynamics and PK/PD Profile of Multiple Subcutaneous Injection of KN057 in Male Patients with Severe Hemophilia a or Moderate-to-Severe Hemophilia B with or Without Inhibitors
Brief Title: KN057 Multiple Dose Study in Patients with Hemophilia a or Hemophilia B with or Without Inhibitors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Alphamab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN057-A-202
Record Dates: First submitted 2024-12-11; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Hemophilia a and B
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- KN057 (Experimental)
  Interventions: Drug: KN057

INTERVENTIONS:
Drug: KN057 — KN057 will be administered subcutaneously once a week.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of KN057 in adult patients with severe Hemophilia A (coagulation factor FVIII activity <1%) or moderate-to-severe Hemophilia B (FIX activity ≤2%). Participants will be administered subcutaneously with KN057 once a week for 20 weeks. KN057 works differently than factor replacement products and will work in the presence of inhibitors. The potential for once weekly subcutaneous administration provides better convenience and compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18-70 years old (including thresholds), body weight ≥40 kg and BMI <30 kg/m^2.
2. Severe Hemophilia A or moderate-to-severe Hemophilia B (coagulation factor FVIII activity <1% or FIX activity ≤2%).
3. Have ≥ 6 treated bleeding episodes within 24 weeks prior to screening (spontaneous and/or traumatic, excluding bleeding episodes related to surgery or traumatic operation).
4. Patients without inhibitors must meet the following criteria: FVIII or FIX inhibitor test is negative during the screening period. Use coagulation factor replacement therapy for no less than 100 exposure days before screening.
5. Patients with inhibitors must meet the following criteria: FVIII or FIX inhibitor test is positive during the screening period. Inhibitors level with high titer positive (≥5 BU/ml) or current low titer positive (<5 BU/ml) refractory to FVIII or FIX replacement and with FVIII or FIX recovery < 60% of expected within previous 12 months prior to screening.

Exclusion Criteria:

1. Those with serious or poorly controlled chronic diseases or obvious systemic diseases: such as cardiovascular system, respiratory system, endocrine and metabolic system, urinary system, digestive system, autoimmune diseases, neurological diseases or psychiatric diseases, bacterial or viral infection, etc.; have previously received lipid-lowering therapy for hypertriglyceridemia or are currently receiving lipid-lowering therapy for hypertriglyceridemia.
2. Have a history of other hereditary or acquired bleeding disorders other than Hemophilia A and Hemophilia B.
3. Have symptoms and signs related to thromboembolic disease or are receiving thrombolytic/antithrombotic treatment; have a history of coronary atherosclerotic disease, arterial or venous thrombosis, or ischemic disease of important organs.
4. Have high risk factors for thrombosis, including reduced activity of antithrombin III, protein S or protein C.
5. When bleeding occurred in the past, rFVIIa was ineffective and (activated) prothrombin complex concentrate (PCC/aPCC) treatment must be used.
6. Are undergoing or planning to undergo immune tolerance induction therapy.
7. Regular use of immunomodulatory therapy, such as regular infusion of immune globulin or regular use of hormones, is required.
8. Those with allergies; those who are allergic to test drugs/similar drugs or excipients; those with a history of multiple allergies (two categories or more); those with a history of specific reactions, such as being allergic to heparin or having experienced heparin-induced thrombocytopenia.
9. Hematological abnormalities: platelet count ≤ 100 × 10^9 /L; hemoglobin < 100g/L; fibrinogen level < lower limit of normal (LLN); prothrombin time > 1.5 times upper limit of normal (ULN).
10. Abnormal liver and kidney function: alanine aminotransferase and/or aspartate aminotransferase >3 times ULN; lactate dehydrogenase >1.5 times ULN; total bilirubin >1.5 times ULN; serum creatinine, triglyceride > ULN; albumin <0.8 times LLN.
11. Chronic active hepatitis B/C virus (HBV/HCV, HBV-DNA or HCV-RNA quantitative detection indicates viral activity); Human immunodeficiency virus (HIV) antibody positive; syphilis antibody positive; Have received antiviral treatment (only for HBV, HCV, and HIV) in the past 3 month, or have plans to undergo antiviral treatment within 28 weeks after the first dose.
12. Have had major surgery within the past 3 months (determined by the investigator), or have elective surgery planned within 28 weeks after the first dose.
13. Due to treatment needs, anti-fibrinolytic or platelet function-affecting drugs need to be used within 5 days before administration or within 28 weeks after the first administration, including medicines, such as aspirin, COX-1 and non-selective non-steroidal anti-inflammatory drugs (NSAIDs, except for acetaminophen), traditional herbal medicine or health supplements at investigator's discretion.
14. Participated in clinical trials related to coagulation factors and received investigational drug treatment within the past 1 month; participated in any other drug clinical trials and received investigational drug treatment within the past 3 months.
15. Have been vaccinated in the past month, or have a vaccination plan within 28 weeks after the first dose, including inactivated vaccine, live attenuated vaccine, recombinant protein vaccine, recombinant adenovirus vaccine, RNA vaccine, DNA vaccine, etc.
16. Subjects with fertile mates are unable to use effective contraception during the study period and within 3 months after the last dose; effective contraceptive methods include: vasectomy, scientific use of male condoms, etc.
17. Have had treatment of Emicizumab within 6 months prior to screening;
18. Have had any prior treatment of genetic therapy for hemophilia.
19. Those participants who drink heavily or are alcoholic within 24 weeks prior to screening or can't avoid heavy drinking during the trial. Heavy drinking means more than 7 units of alcohol per week, 1 unit=360ml of beer, or 45ml of liquor with 40% alc/vol, or 150ml of wine.
20. Other factors that the investigator considers inappropriate for participation in this trial.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events(TEAEs) | Week 0 up to Week 26
  TEAEs are adverse events occurred following the start of treatment or adverse events increasing in severity during treatment.
Number of participants with abnormal laboratory findings in Hematology | Week 0 up to Week 26
  Including white blood cells, red blood cells, lymphocyte count, neutrophil count, monocyte count, eosinophil count, basophil count, lymphocyte percentage, neutrophil percentage, monocyte percentage, eosinophil percentage, basophil percentage, hemoglobin, hematocrit, platelet count.
Number of participants with abnormal laboratory findings in Coagulation Function | Week 0 up to Week 26
  Including prothrombin time (PT), international normalized ratio (INR), activated partial thrombin time (APTT), thrombin time (TT), fibrinogen (FBG/FIB), D-dimer (D-Di), fibrin(ogen) degradation product (FDP), antithrombin-Ⅲ (AT-Ⅲ)
Number of participants with abnormal laboratory findings in Blood Biochemistry | Week 0 up to Week 26
  Including total bilirubin (TBIL), indirect bilirubin (IBIL), direct bilirubin (DBIL), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), alkaline phosphatase (ALP), total protein (TP), albumin (ALB), globulin, white globulin ratio , urea and/or urea nitrogen (BUN) (collected according to the specific test item at the clinical site), creatinine (Cr), uric acid, glucose, total cholesterol (TC), triglycerides (TG), low-density lipoprotein (LDL), high-density lipoprotein (HDL), lactate dehydrogenase (LDH), creatine kinase, sodium , potassium, chloride, calcium, C- reactive protein.
Number of participants with clinically significant changes in 12-lead electrocardiograms | Week 0 up to Week 26
Number of participants with clinically significant changes in vital signs | Week 0 up to Week 26
  Heart Rate, Respirations, Temperature, Blood Pressure
Number of participants with clinically significant changes in physical examination Findings | Week 0 up to Week 26
Incidence and severity of injection site reaction | Week 0 up to Week 26

SECONDARY OUTCOMES:
Plasma Concentration of KN057 | Week 0 up to Week 26
Maximum Plasma Concentration (Cmax) of KN057 | Week 0 up to Week 26
Time to Reach Maximum Plasma Concentration (Tmax) of KN057 | Week 0 up to Week 26
Maximum observed KN057 concentration at steady-state | Week 0 up to Week 26
Area Under the Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of KN057 | Week 0 up to Week 26
Apparent Clearance (CL/F) of KN057 | Week 0 up to Week 26
Changes of Free Tissue factor pathway inhibitor (TFPI) from baseline | Week 0 up to Week 26
  Tissue factor pathway inhibitor (TFPI) is an anticoagulant protein that inhibits early phases of the procoagulant response.
Changes of Total TFPI from baseline | Week 0 up to Week 26
  TFPI: Tissue factor pathway inhibitor
Changes of Prothrombin fragment 1+2 (PF1+2) from baseline | Week 0 up to Week 26
The number and proportion of participants who produce anti-KN057 antibody | Week 0 up to Week 26
The number and proportion of participants who produce anti-KN057 neutralizing antibodies | Week 0 up to Week 26
Annualized Bleeding Rate (ABR) | Week 0 up to Week 20
  ABR=number of bleeding episodes reported in visit days÷visit days×365.25

IPD SHARING:
Plan to Share IPD: Undecided